CLINICAL TRIAL: NCT02491255
Title: REPRISE Japan: Repositionable Percutaneous Replacement of Stenotic Aortic Valve Through Implantation of Lotus™ Valve System - Clinical Evaluation in Japan
Brief Title: Safety and Efficacy Study of Lotus Valve for Transcatheter Aortic Valve Replacement (REPRISE Japan)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S6002
Record Dates: First submitted 2015-06-18; First posted 2015-07-08 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lotus Valve System (Experimental): Transcatheter aortic valve replacement (TAVR) with Lotus Valve System
  Interventions: Device: Lotus Valve System

INTERVENTIONS:
Device: Lotus Valve System — Device: Lotus Valve System

SUMMARY:
The objective of this study is to confirm the safety and effectiveness of the Lotus™ Valve System in the Japanese medical environment for transcatheter aortic valve replacement (TAVR) in symptomatic subjects with calcific, severe native aortic stenosis who are considered at high or extreme risk for surgical valve replacement.

DETAILED DESCRIPTION:
A prospective, multicenter trial designed to confirm that the safety and effectiveness of the Lotus Valve System in the Japanese medical environment are consistent with the REPRISE III results for TAVR in symptomatic subjects who have calcific, severe native aortic stenosis and who are at extreme or high risk for surgical valve replacement.

ELIGIBILITY:
IC1. Subject has documented calcific, severe native aortic stenosis with an initial AVA of ≤1.0 cm2 (or AVA index of ≤0.6 cm2/m2) and a mean pressure gradient ≥40 mm Hg or jet velocity ≥4.0 m/s, as measured by echocardiography and/or invasive hemodynamics.

IC2. Subject has a documented aortic annulus size of ≥18 mm and ≤27 mm based on the Center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]) and is deemed treatable with an available size of the test device

IC3. Subject has symptomatic aortic valve stenosis with NYHA Functional Class ≥ II

IC4. There is agreement by the heart team (which must include a site investigator interventionalist and a site investigator cardiac surgeon) that subject is at high or extreme operative risk for surgical valve replacement (see note below for definitions of extreme and high risk, the required level of surgical assessment, and CRC confirmation) and that TAVR is appropriate. Additionally, subject has at least one of the following.

* Society of Thoracic Surgeons (STS) score ≥8% -OR-
* If STS <8, subject has at least one of the following conditions:

  * Hostile chest
  * Porcelain aorta
  * Severe pulmonary hypertension (>60 mmHg)
  * Prior chest radiation therapy
  * Coronary artery bypass graft(s) at risk with re-operation
  * Severe lung disease (need for supplemental oxygen, FEV1 <50% of predicted, DLCO <60%, or other evidence of severe pulmonary dysfunction)
  * Neuromuscular disease that creates risk for mechanical ventilation or rehabilitation after surgical aortic valve replacement
  * Orthopedic disease that creates risk for rehabilitation after surgical aortic valve replacement
  * Childs Class A or B liver disease (subjects with Childs Class C disease are not eligible for inclusion in this trial)
  * Frailty as indicated by at least one of the following: 5-meter walk >6 seconds, Katz ADL score of 3/6 or less, body mass index <21, wheelchair bound, unable to live independently
  * Age ≥90 years
  * Other evidence that subject is at high or extreme risk for surgical valve replacement (CRC must confirm agreement with site heart team that subject meets high or extreme risk definition)

IC5. Heart team (which must include a cardiac interventionalist and an experienced cardiac surgeon) assessment that the subject is likely to benefit from valve replacement.

IC6. Subject (or legal representative) understands the study requirements and the treatment procedures, and provides written informed consent.

IC7. Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.

IC8. Subject must be at least 20 years old.

IC9. For subjects not suitable for iliofemoral access (because of caliber of the iliofemoral vessels, severe tortuosity or other factors preventing safe iliofemoral access), trans-aortic access is deemed appropriate by the heart team and confirmed by the CRC. This inclusion criterion is only applicable to the TAo substudy and the 21mm substudy if the transaortic approach is used.

Note: Extreme operative risk and high operative risk are defined as follows:

Extreme Operative Risk: Predicted operative mortality or serious, irreversible morbidity risk ≥50% at 30 days.

High Operative Risk: Predicted operative mortality or serious, irreversible morbidity risk ≥15% at 30 days.

EC1. Subject has a congenital unicuspid or bicuspid aortic valve.

EC2. Subject has had an acute myocardial infarction within 30 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK-MB elevation and/or troponin elevation).

EC3. Subject has had a cerebrovascular accident or transient ischemic attack within the past 6 months prior to study enrollment.

EC4. Subject has end-stage renal disease or has eGFR <20. Note: eGFR(ml/min/1.73m2)=194×Cr-1.094×Age-0.287×(If female×0.739)

EC5. Subject has a pre-existing prosthetic aortic or mitral valve.

EC6. Subject has severe aortic, tricuspid, or mitral regurgitation.

EC7. Subject has a need for emergency surgery for any reason.

EC8. Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.

EC9. Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.

EC10. Subject has Hgb <9 g/dL, platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.

EC11. Subject requires chronic anticoagulation therapy after the implant procedure and cannot be treated with warfarin (other anticoagulants are not permitted in the first month) for at least 1 month concomitant with either aspirin or P2Y12 inhibitor (clopidogrel or ticlopidine, but prasugrel is not allowed).

EC12. Subject had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months, or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen, or will refuse transfusions.

EC13. Subject has known hypersensitivity to contrast agents that cannot be adequately pre-medicated, or has known hypersensitivity to aspirin, all P2Y12 inhibitors, heparin, nickel, tantalum, titanium, or polyurethanes.

EC14. Subject has a life expectancy of less than 12 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment.

EC15. Subject has hypertrophic obstructive cardiomyopathy.

EC16. Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty or pacemaker implantation, which are allowed).

EC17. Subject has untreated coronary artery disease, which in the opinion of the treating physician is clinically significant and requires revascularization.

EC18. Subject has severe left ventricular dysfunction with ejection fraction <20%.

EC19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.

EC20. Subject has severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely, marked tortuosity, significant narrowing of the abdominal aorta, severe unfolding of the thoracic aorta, or symptomatic carotid or vertebral disease). This exclusion criterion is only applicable to the TF study and the 21mm substudy if the transfemoral or transiliac approach is used.

EC21. Subject has thick (>5 mm) protruding or ulcerated atheroma in the aortic arch. This exclusion criterion is only applicable to the TF study and the 21mm substudy if the transfemoral or transiliac approach is used.

EC22. Subject has arterial access that is not acceptable for the test device delivery systems as defined in the device Instructions For Use.

EC23. Subject has current problems with substance abuse (e.g., alcohol, etc.).

EC24. Subject is participating in another investigational drug or device study that has not reached its primary endpoint.

EC25. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation. Enrollment is permissible after permanent pacemaker implantation.

EC26. Subject has severe incapacitating dementia.

EC27. Subject is a woman who is pregnant, nursing (a pregnancy test must be performed in women of potential child-bearing) or wishes to be pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint: Composite of all-cause mortality, stroke, life-threatening and major bleeding events, stage 2 or 3 acute kidney injury, or major vascular complications | 30 days following procedure
Primary Effectiveness Endpoint: Composite of all-cause mortality, disabling stroke(adjudicated by an independent CEC), or moderate or greater paravalvular aortic regurgitation(based on independent core laboratory assessment) | 6 month following procedure

SECONDARY OUTCOMES:
Moderate or greater paravalvular aortic regurgitation (based on core lab assessment) | 6 month following procedure

OTHER OUTCOMES:
Successful deployment of the study valve | at discharge or 7 days post-procedure (whichever comes first)
Successful retrieval of the study valve if retrieval is attempted | at discharge or 7 days post-procedure (whichever comes first)
Successful repositioning of the study valve if repositioning is attempted | at discharge or 7 days post-procedure (whichever comes first)
Grade of aortic valve regurgitation: paravalvular, central, and combined | at discharge or 7 days post-procedure (whichever comes first)
Clinical procedural success | 30 days post procedure
  Defined as implantation of the test device in the absence of death, disabling stroke, major vascular complications, and life-threatening or major bleeding
Procedural success | 30 days post procedure
  defined as absence of procedural mortality, correct positioning of a single transcatheter valve into the proper anatomical location , intended performance of the study device at 30 days (effective orifice area [EOA] >0.9 cm2 for body surface area (BSA) <1.6 m2 and EOA >1.1 cm2 for BSA ≥1.6 m2 plus either a mean aortic valve gradient <20 mm Hg or a peak velocity <3m/sec, and no moderate or severe prosthetic valve aortic regurgitation) plus no serious adverse events
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | At discharge or 7 days post-procedure (whichever comes first)
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 30 days post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 6 months post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 1 year post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 2 years post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 3 years post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 4 years post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Additional indications of prosthetic aortic valve performance as measured by transthoracic echocardiography | 5 years post procedure
  assessed by an independent core laboratory, including effective orifice area, mean and peak aortic gradients, peak aortic velocity, and grade of aortic regurgitation
Health status as evaluated by Quality of Life questionnaires | baseline, 1 and 6 months; and 1, 3, and 5 years
  SF-12 and Kansas City Cardiomyopathy
Mortality: all-cause, cardiovascular, and non-cardiovascular | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Stroke: disabling and non-disabling | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Myocardial infarction (MI): periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Bleeding: life-threatening (or disabling) and major | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Acute kidney injury based on the AKIN System Stage 3 (including renal replacement therapy) or Stage 2 | ≤7 days post index procedure
Major vascular complication | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Repeat procedure for valve-related dysfunction (surgical or interventional therapy) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
Hospitalization for valve-related symptoms or worsening congestive heart failure (New York Hear Association [NYHA] class III or IV) | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
New permanent pacemaker implantation resulting from new or worsened conduction disturbances | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post procedure
New onset of atrial fibrillation or atrial flutter | Within the index hospitalization
Coronary obstruction | ≤72 hours post index procedure
Ventricular septal perforation | ≤72 hours post index procedure
Mitral apparatus damage | ≤72 hours post index procedure
Cardiac tamponade | ≤72 hours post index procedure
Prosthetic aortic valve malpositioning, including valve migration, valve embolization, or ectopic valve deployment | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post index procedure
Transcatheter aortic valve (TAV)-in-TAV deployment | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post index procedure
Prosthetic aortic valve thrombosis | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post index procedure
Prosthetic aortic valve endocarditis | At discharge or 7 days post-procedure (whichever comes first), 30 days, 6 months, and 1, 2, 3, 4, and 5 years post index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiki Sawa, Principal Investigator — Osaka University Hospital; Shigeru Saito, Principal Investigator — Shonankamakura General Hospital
Locations (5):
- Japan (5):
  - Shonankamakura General Hospital, Kamakura, Kanagawa
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Osaka University Hospital, Suita, Osaka
  - Sakakibara Heart Institute, Fuchū, Tokyo
  - Keio University Hospital, Shinjuku, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided